CLINICAL TRIAL: NCT06039228
Title: Thriving Through the Storms: A School-based Mental Health Promotion Program for Building Psychological Flexibility and Resilience
Brief Title: School-based Group Acceptance and Commitment Therapy for Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Jennifer Yee Man Tang, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KPF23GWP12
Record Dates: First submitted 2023-09-09; First posted 2023-09-15 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Depressive Symptoms; Anxiety; Stress
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Behavioral: Acceptance and commitment therapy

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy — Four sessions of group acceptance and commitment therapy, with each session lasting for 1.5 hours.

SUMMARY:
The objective of the investigators' mental health promotion intervention premised on the Acceptance and Commitment Therapy (ACT) framework in secondary school settings aims to enhance young people's psychological flexibility and reduce their emotional distress. ACT is an evidence-based approach that encourages individuals to act in alignment with their identified values. The investigator's team will employ an ACT protocol for adolescents developed by Louise Hayes and Joseph Ciarrochi. The study includes a single-group study design. The investigator will compare the pre- and post-intervention data to assess the feasibility and potential effectiveness of the group intervention.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants are adolescents who reported mild to moderate severity of psychological distress, including those who report:

* a score of 5-19 on the Patient Health Questionnaire (PHQ-9), or
* a score of 5-14 on the General Anxiety Disorder-7, or
* a score ≥14 on the Perceived Stress Scale.

Exclusion Criteria:

Adolescents will be excluded if they exhibit or report:

* violent or aggressive behavior, or
* active self-injurious or suicidal thought, or
* active psychotic symptom.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Acceptance and Action Questionnaire - II | Baseline and 4 weeks
The 14-item Resilience Scale | Baseline and 4 weeks
Patient Health Questionnaire - 9 | Baseline and 4 weeks
General Anxiety Disorder - 7 | Baseline and 4 weeks
Perceived Stress Scale | Baseline and 4 weeks

SECONDARY OUTCOMES:
Satisfaction with Life Scale | Baseline and 4 weeks
Pittsburgh Sleep Quality Index | Baseline and 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Educational Psychology, The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No